CLINICAL TRIAL: NCT03458702
Title: The Effects of Yoga and Quiet Rest on Subjective Levels of Anxiety and Physiological Correlates: A 2-way Randomized Crossover Design
Brief Title: The Effects of Emotional Exposure on State Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 504055
Record Dates: First submitted 2018-02-16; First posted 2018-03-08 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: autonomic function; emotion; heart rate variability
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Methods: A randomized repeated-measures crossover clinical trial was performed. Forty healthy, female college students completed a 30 min session of YogaFit and a time-matched seated rest condition on separate days. After each condition, participants viewed 30 min of emotional picture stimuli. State anxiety, heart rate and time-domain and frequency-domain measures of HRV were assessed baseline, post- condition, and post-exposure to emotional stimuli.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YogaFit then Quiet Rest (Experimental): Participants participated in a 30 min YogaFit and then a session of 30 min of Quiet Rest on a separate day.
  Interventions: Behavioral: YogaFit; Behavioral: Quiet Rest
- Quiet Rest then YogaFit (Experimental): Participants participated in a 30 min Quiet Rest session and then a session of 30 min of YogaFit on a separate day.
  Interventions: Behavioral: YogaFit; Behavioral: Quiet Rest

INTERVENTIONS:
Behavioral: YogaFit — For YogaFit Vinyasa Flow (referred to as YogaFit in this manuscript)], participants followed, via digital versatile disc, a standardized YogaFit format choreographed by an American Council of Exercise Certified and Registered Yoga Teacher (RYT). YogaFit was performed in the same laboratory setting and lasted 30 min. YogaFit is a westernized version of yoga that does not use Sanskrit terms (Shaw 2009). Breath was an integral part of every movement with specific breath rates for each phase of the session. The objective was to move the body with intention and purpose and be present in the body.
Behavioral: Quiet Rest — Participants completed 30 min of quiet rest

SUMMARY:
A randomized repeated-measures crossover clinical trial was performed. Forty healthy, female college students completed a 30 min session of YogaFit and a time-matched seated rest condition on separate days. After each condition, participants viewed 30 min of emotional picture stimuli. State anxiety, heart rate and time-domain and frequency-domain measures of HRV were assessed baseline, post- condition, and post-exposure to emotional stimuli. Data were analysed using a condition x time (2 × 3) repeated-measures ANOVA.

DETAILED DESCRIPTION:
The design was a repeated-measures randomized crossover trial. Each study participant completed 4 different sessions on 4 different days: (day 1) participant screening; (day 2 or 3) study condition A (seated, quiet rest); (alternate day 2 or 3) study condition B (moderate-intensity YogaFit); and (day 4) a session to rate IAPS pictures (14) and undergo a single DEXA scan [Prodigy/301776R. G.E. Medical Systems-Lunar DEXA Scanner, Fairfield, CT, USA]. Utilizing a simple randomization process, participants were randomized in a 1:1 ratio to participate in either the YogaFit condition or the quiet rest condition. The study conditions were counterbalanced and alternated using odd and even numbers to begin the sequence. Participants were not informed if the first condition was A or B. Self-reported anxiety levels and 10 min of continuous physiological data were collected: (a) baseline; (b) post-condition; and (c) post-exposure for both condition A and B. All participants completed both the psychological and physiological assessments. Both experimental conditions A and B were completed in 90 min. To ensure compliance, participants were observed through a glass window every 10 min during study conditions. Testing time and procedures were identical with the exception of the experimental condition on days two and three.

All participants were familiarized with the videotaped YogaFit session before participating in the study. Participants were instructed to arrive for all visits dressed in loose fitting athletic wear and were asked to refrain from all food, alcohol, caffeine, gum chewing or the use of tobacco products 3 h before their scheduled meeting in the laboratory.

During pre-screening, participants completed: (a) a standard health history questionnaire; (b) the STAI-Y2; (c) the BDI and (d) a custom DEXA safety questionnaire. Qualified participants were then asked to track their menstrual cycle using a menstrual log and e-mail the primary investigator on day 1 of the follicular phase of their menstrual cycle, thus using the first day of the women's menstrual cycle to generate an unpredictable random sequence and to eliminate any sequence bias. The participant was then scheduled for condition A first or condition B first. The conditions were counterbalanced to control for order effects, with odd numbers beginning condition A first and even numbers beginning condition B first. To control for the effects of the menstrual cycle on anxiety, participants completed condition A and condition B within a 7-day period during the follicular phase of their menstrual cycle (specifically days 1-10). Participants were also asked to maintain pre-study physical activity levels during the 7-day period. All testing was completed by day 10 of their menstrual cycle. State anxiety was psychologically quantified using a reliable and validated assessment of anxiety, Spielberger's State-Trait Anxiety Inventory (STAI-YI).

Instruments for testing all physiological variables were calibrated and used by the same investigator in order to control possible inter-tester variation. During both condition A and B, a ProComp Infiniti System with Biograph software version 6.0 was used to measure HR and indices of HRV at a sampling rate of 2048 cycles per sec at the 3 different time points. Three electrodes were placed on the participants to monitor HR as specified by the ProComp Infiniti System. The negative electrode was placed in the right shoulder fossa below the clavicle, the positive electrode was placed medially on the thorax below the sternum, and the ground electrode was placed in the left shoulder fossa below the clavicle. Indices of HRV included the time-domain variable, root mean square of successive differences (RMSSD) and two frequency-domains: the low frequency power bands and the high frequency power bands in normalized units (LFNU and HFNU, respectively).

Measures of HR and HRV were analysed using CardioPro Infinity-HRV Analysis Software Module-SA7J90 [ProComp Infiniti System, Montreal, Quebec, Canada: Cimetra LLC]. An accelerometer using the ActiLife 6 Software and a Polar Heart Rate Sensor were strapped to the participant and used to monitor the intensity level of both study conditions A and B. The accelerometer was used only to record HR data and no other accelerometer data were analysed. Participants were then informed of the experimental condition. For study condition A (quiet, seated rest), participants sat on a yoga mat in a cross-legged position for 30 min in a quiet laboratory setting. For study condition B [YogaFit Vinyasa Flow (referred to as YogaFit in this manuscript)], participants followed, via digital versatile disc, a standardized YogaFit format choreographed by a certified American Council of Exercise Instructor and Registered Yoga Alliance Teacher. Yoga- Fit was performed in the same laboratory setting and lasted 30 min. There are 7 principles of alignment that are applied in every YogaFit session: (1) establish a base and dynamic tension; (2) create core stability; (3) align the spine; (4) soften and align the knees; (5) relax shoulders back and down; (6) hinge at the hips; and (7) shorten the lever. The YogaFit essence is based on: Breathing, Feeling, Listening to the Body, Letting Go of Competition, Judgement, Expectations, and Staying in the Present Moment. The movements included in each specific phase were chosen from Beth Shaw's YogaFit Vinyasa Flow Series. To measure intensity of theYogaFit routine, ratings of perceived exertion (RPE) [24] were recorded following both condition A and B. The accelerometer and heart rate sensor were removed after the study condition. After both study conditions, participants again completed STAI-Y1 and 10 min of post-condition data were collected. Participants then viewed 90 emotionally arousing pictures from the IAPS after both study conditions A and B. Pictures were viewed on a 70" × 70"portable projection screen. The 90 pictures were arranged in 3 blocks of 30; each block contained 10 pictures from each valence category. Among the 90 pictures used, 30 were pleasant (15 erotica and 15 babies, families, and cute animals); 30 were neutral (15 neutral people and 15 neutral objects and scenes); and 30 were unpleasant (15 threat and 15 mutilation) based on normative ratings of valence [5]. No more than two pictures from the same category appeared consecutively. Two different picture orders were constructed and counterbalanced across testing day and experimental condition. Each picture was shown for 4-s, followed by a 12-, 14-, or 16-s inter-picture interval, which consisted of a centrally located fixation cross. The total picture-viewing time, including brief breaks between each picture block, was approximately 30 min. Participants were instructed to look at each picture the entire time it was on the monitor and to subjectively categorize each picture as pleasant, neutral, or unpleasant using a response pad [E-Prime 2.0, Psychology Software Tools, Inc., Pittsburgh, PA, USA] resting on their lap. These ratings were not used to compare to the normative ratings, but rather, the purpose of categorizing the pictures was to ensure that participants concentrated on the pictures. Immediately after viewing the pictures, participants again completed STAI-Y1 and 10 min post-exposure data were collected. In accordance with the Center for the Study of Emotion and Attention, participants were also asked to rate the IAPS images in order to further image standardization. Participants rated each of the 90 pictures (hard copy, one picture per page in a standard, self-paced order) using the Self-Assessment Manikin (SAM) during visit 4 to the laboratory. Additionally, participants underwent a single DEXA scan for body composition assessment.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria included women who:

* were between 18 and 25 years of age;
* were not suffering from any medical conditions that would influence the results or compromise safety during training-such as disorders effecting balance, or pregnancy;
* who were not taking antidepressant or anti-anxiety medication;
* were not clinically diagnosed with generalized anxiety disorder in the previous six months;
* were within the normal range (± 1 SD from the M) for female college students for trait anxiety according to Spielberger's Trait Anxiety Inventory [(STAI-Y2); range: 40.40 ± 10.15] (Spielberger 1983);
* were within normal (minimal to mild) levels of depression according to the Beck Depression Inventory [(BDI); range: 0-18] (Oliver and Simmons 1984);
* had a normal menstrual cycle (cycles occurring less than every 26 to 35 days and lasting less than 2 or more than 7 days);
* were not considered high-risk for dual energy x-ray absorptiometry (DEXA) based on a standardized questionnaire approved by the University Radiation Safety Committee; and
* were familiar with yoga or had not participated in at least 3 yoga practice sessions.

Exclusion Criteria:

* The exclusion criteria included women who:

  * were less than 18 or more than 25 years of age;
  * were suffering from any medical conditions that would influence the results or compromise safety during training-such as disorders effecting balance, or pregnancy;
  * who were taking antidepressant or anti-anxiety medication;
  * were clinically diagnosed with generalized anxiety disorder in the previous six months;
  * were not within the normal range (± 1 SD from the M) for female college students for trait anxiety according to Spielberger's Trait Anxiety Inventory [(STAI-Y2); range: 40.40 ± 10.15];
  * were not within normal (minimal to mild) levels of depression according to the Beck Depression Inventory [(BDI); range: 0-18];
  * had an abnormal menstrual cycle (cycles occurring less than every 26 to 35 days and lasting less than 2 or more than 7 days);
  * were considered high-risk for dual energy x-ray absorptiometry (DEXA) based on a standardized questionnaire approved by the University Radiation Safety Committee; and
  * were not familiar with yoga or had not participated in at least 3 yoga practice sessions.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2014-03-15 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacalyn Robert-McComb, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albracht-Schulte K, Robert-McComb J. The effects of yoga and quiet rest on subjective levels of anxiety and physiological correlates: a 2-way crossover randomized trial. BMC Complement Altern Med. 2018 Oct 17;18(1):280. doi: 10.1186/s12906-018-2343-1. PMID 30333014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited women from yoga classes at the university.
Pre-assignment Details: Qualified participants were asked to track their menstrual cycle using a menstrual log and e-mail the primary investigator on day 1 of the follicular phase of their menstrual cycle. The participant was then scheduled for condition A first or condition B first.
Groups:
- YogaFit Then Quit Rest: Participants completed a 30 min YogaFit Session and then a 30 min Quiet Rest Session on different days.
  YogaFit: For YogaFit Vinyasa Flow (referred to as YogaFit in this manuscript)], participants followed, via digital versatile disc, a standardized YogaFit format choreographed by an American Council of Exercise Certified and Registered Yoga Teacher (RYT). YogaFit was performed in the same laboratory setting and lasted 30 min. YogaFit is a westernized version of yoga that does not use Sanskrit terms (Shaw 2009). Breath was an integral part of every movement with specific breath rates for each phase of the session. The objective was to move the body with intention and purpose and be present in the body.
  On another day, participants completed 30 min of Quiet Rest
- Quiet Rest Then Yoga Fit: Participants completed 30 min of Quiet Rest and then 30 min of YogaFit on different days.
Period: Study Condition A (Yoga or Rest)
Arm/Group | YogaFit Then Quit Rest | Quiet Rest Then Yoga Fit
Started | 28 | 28
Completed | 24 | 22
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 4 | 6
Period: Study Condition B (Yoga or Rest)
Arm/Group | YogaFit Then Quit Rest | Quiet Rest Then Yoga Fit
Started | 24 | 22
Completed | 20 | 20
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2
Period: Picture Rating/Body Composition
Arm/Group | YogaFit Then Quit Rest | Quiet Rest Then Yoga Fit
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- YogaFit and Quit Rest: Participants completed 30 min of YogaFit and then 30 min of Quiet Rest on different days.
  YogaFit: For YogaFit Vinyasa Flow (referred to as YogaFit in this manuscript)], participants followed, via digital versatile disc, a standardized YogaFit format choreographed by an American Council of Exercise Certified and Registered Yoga Teacher (RYT). YogaFit was performed in the same laboratory setting and lasted 30 min. YogaFit is a westernized version of yoga that does not use Sanskrit terms (Shaw 2009). Breath was an integral part of every movement with specific breath rates for each phase of the session. The objective was to move the body with intention and purpose and be present in the body.
Arm/Group | YogaFit and Quit Rest
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
STAI-Y2 score [Mean (Standard Deviation); unit: units on a scale] — This is Spielberger's Trait Anxiety Score. Range = 20-80. Higher scores indicate increased trait anxiety.
  units on a scale | 39.05 (5.91)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — This is the score from the Back Depression Inventory. Scores range 0-63. Higher scores indicate increased depression.
  units on a scale | 7.68 (4.21)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — The BMI is computed by this formula kg/m2. BMI < 18.5 = underweight, BMI =18.5 - 24.9 = normal weight, BMI = 25 - 29.9 = overweight, BMI > 30 = obese
  kg/m^2 | 23.21 (3.12)
Body Fat Percentage [Mean (Standard Deviation); unit: percentage] — DEXA was used to calculate body fat percentage.
  percentage | 34.94 (7.58)

OUTCOME MEASURES:

1. Primary Outcome: STAI-Y1 Score Assessed at Baseline, Post-Condition and Post-Exposure
Description: State anxiety (STAI-Y1 score) at baseline ( 10 min prior to condition), post-condition (10 min after completion of YogaFit and Quiet Rest) and post-exposure (10 min after completion of 30 min of viewing emotional pictures from the International Affective Picture System (IAPS)) was measured by Spielberger's 20 question State Anxiety Questionnaire (STAI-YI). Scores range from 20-80, with higher scores indicative of increased state anxiety.
Time Frame: 10 min prior to condition, 10 min after completion of YogaFit and Quiet Rest,10 min after exposure to emotional stimuli
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Quiet Rest: 30 min of Quiet Rest
Arm/Group | YogaFit | Quiet Rest
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 33.48 (9.41) | 33.53 (10.63)
  Post-Condition | 27.43 (7.05) | 29.78 (7.82)
  Post-Exposure | 33.18 (10.75) | 34.48 (10.34)
Statistical Analysis 1: Comparison: YogaFit vs Quiet Rest; Test type: Equivalence — It would be expected at baseline that there were no differences between groups; p > .05, t-test, 2 sided
Statistical Analysis 2: Comparison: YogaFit vs Quiet Rest; ANOVA for TIME; Test type: Superiority; p < 0.001, ANOVA

2. Primary Outcome: Heart Rate Assessed at Baseline, During Condition, Post-Condition and Post-Exposure
Description: HR in beats per min assessed utilizing three electrodes and ProComp Infiniti Software at baseline (10 min prior to condition), during the condition (30 min of YogaFit and Quiet Rest), post-condition (10 min after YogaFit and Quiet Rest) and post-exposure (10 min after 30 min of viewing emotional pictures from the International Affective Picture System (IAPS)).
Time Frame: 10 min prior to condition, 30 min during condition, 10 min after completion of YogaFit and Quiet Rest,10 min after exposure to emotional stimuli
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | YogaFit | Quiet Rest
Number analyzed (Participants) | 40 | 40
beats per minute
  Baseline | 72.48 (10.61) | 73.59 (11.25)
  During Condition | 101.01 (22.65) | 69.35 (10.61)
  Post-Condition | 74.51 (10.39) | 70.43 (9.77)
  Post-Exposure | 71.69 (9.73) | 70.17 (9.65)
Statistical Analysis 1: Comparison: YogaFit vs Quiet Rest; Test type: Equivalence — It would be expected at baseline there would be no difference between groups; p > .05, ANOVA
Statistical Analysis 2: Comparison: YogaFit vs Quiet Rest; ANOVA: Condition x Time Interaction; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: YogaFit vs Quiet Rest; ANOVA: TIME; Test type: Superiority; p = 0.005, ANOVA

3. Primary Outcome: Root Mean Square of Successive Differences (RMSSD) Assessed at Baseline, Post-Condition and Post-Exposure
Description: A measure of HRV, RMSSD, was assessed using three electrodes and CardioPro Infiniti-HRV Analysis Software at baseline (10 min prior to condition), post-condition (10 min after completion of YogaFit and Quiet Rest) and post-exposure (10 min after 30 min of viewing emotional pictures from the International Affective Picture System (IAPS)). HRV is associated with good health: increased RMSSD is thought to be beneficial.
Time Frame: 10 min prior to condition, 10 min after completion of YogaFit and Quiet Rest,10 min after exposure to emotional stimuli
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | YogaFit | Quiet Rest
Number analyzed (Participants) | 40 | 40
milliseconds
  Baseline | 61.32 (30.80) | 61.87 (33.98)
  Post-Condition | 62.41 (36.33) | 75.66 (40.67)
  Post-Exposure | 72.75 (43.11) | 79.41 (42.49)
Statistical Analysis 1: Comparison: YogaFit vs Quiet Rest; Test type: Equivalence — It would be hypothesized that there would not be a difference at baseline; p > .05, ANOVA
Statistical Analysis 2: Comparison: YogaFit vs Quiet Rest; ANOVA: CONDITION X TIME INTERACTION; Test type: Superiority; p = 0.042, ANOVA
Statistical Analysis 3: Comparison: YogaFit vs Quiet Rest; ANOVA: TIME; Test type: Superiority; p < 0.001, Chi-squared, Corrected

4. Primary Outcome: Low-frequency Band (LFNU) Assessed at Baseline, Post-Condition and Post-Exposure
Description: A measure of HRV, LFNU, assessed using three electrodes and CardioPro software at baseline (10 min prior to condition), post-condition (10 min after YogaFit and Quiet Rest) and post-exposure (10 min after 30 min of viewing emotional pictures from the International Affective Picture System (IAPS)).
  Low frequency (LF) is defined as 0.04-0.15 Hz (cycles per s) or a band ranging from 0.04 Hz to 0.15 Hz. High frequency (HF) is defined as a band ranging from 0.15-0.4 Hz (cycles per s). The most common frequency domain parameters include the powers in absolute and relative terms and the normalized power of the HF and LF bands or expressed as normalized units.
  The formula for n.u. for LF = LF in ms2/LF in ms2 + LF in ms2
  HRV is associated with good health: increased LFNU is thought to be beneficial.
Time Frame: 10 min prior to condition, 10 min after completion of YogaFit and Quiet Rest,10 min after exposure to emotional stimuli
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | YogaFit | Quiet Rest
Number analyzed (Participants) | 40 | 40
ratio
  Baseline | 53.50 (17.13) | 53.75 (17.93)
  Post-Condition | 52.56 (16.07) | 54.50 (17.77)
  Post-Exposure | 58.42 (13.86) | 56.52 (15.18)
Statistical Analysis 1: Comparison: YogaFit vs Quiet Rest; Test type: Equivalence — A difference at baseline was not expected; p > .05, ANOVA
Statistical Analysis 2: Comparison: YogaFit vs Quiet Rest; ANOVA: TIME; Test type: Superiority; p = 0.016, ANOVA

5. Primary Outcome: High-frequency Band (HFNU) Assessed at Baseline, Post-Condition and Post-Exposure
Description: A measure of HRV, HFNU, assessed using three electrodes and CardioPro software at baseline (10 min prior to condition), post-condition (10 min after completion of YogaFit and Quiet Rest) and post-exposure (10 min after 30 min of viewing emotional pictures from the International Affective Picture System (IAPS)).
  High frequency (HF) is defined as a band ranging from 0.15-0.4 Hz (cycles per s). Low frequency (LF) is defined as 0.04-0.15 Hz (cycles per s) or a band ranging from 0.04 Hz to 0.15 Hz. The most common frequency domain parameters include the powers in absolute and relative terms and the normalized power of the HF and LF bands or expressed as normalized units. The formula for n.u. for HF = HF in ms2/LF in ms2 + LF in ms2.
  HRV is associated with good health: HFNU and LFNU are negatively correlated.
Time Frame: 10 min prior to condition, 10 min after completion of YogaFit and Quiet Rest,10 min after exposure to emotional stimuli
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | YogaFit | Quiet Rest
Number analyzed (Participants) | 40 | 40
ratio
  Baseline | 46.49 (17.13) | 46.25 (17.93)
  Post-Condition | 47.19 (16.22) | 44.55 (17.89)
  Post-Exposure | 41.58 (13.86) | 43.55 (15.15)
Statistical Analysis 1: Comparison: YogaFit vs Quiet Rest; Test type: Equivalence — no difference is expected at baseline; p > .05, ANOVA
Statistical Analysis 2: Comparison: YogaFit vs Quiet Rest; ANOVA:TIME; Test type: Superiority; p = 0.026, ANOVA

6. Secondary Outcome: RPE Assessed Post-Condition
Description: Ratings of perceived exertion (RPE) assessed using Borg's scale of perceived exertion and pain. Scores range from 6-20, with 6 indicating no exertion at all.
Time Frame: Post-Condition, 10 min after completion of YogaFit and Quiet Rest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | YogaFit | Quiet Rest
Number analyzed (Participants) | 40 | 40
score on a scale | 10.83 (1.66) | 6.05 (0.22)
Statistical Analysis 1: Comparison: YogaFit vs Quiet Rest; Test type: Superiority; p < .05, t-test, 1 sided

ADVERSE EVENTS:
Groups:
- YogaFit: Participants completed a 30 min YogaFit Session.
  YogaFit: For YogaFit Vinyasa Flow (referred to as YogaFit in this manuscript)], participants followed, via digital versatile disc, a standardized YogaFit format choreographed by an American Council of Exercise Certified and Registered Yoga Teacher (RYT). YogaFit was performed in the same laboratory setting and lasted 30 min. YogaFit is a westernized version of yoga that does not use Sanskrit terms (Shaw 2009). Breath was an integral part of every movement with specific breath rates for each phase of the session. The objective was to move the body with intention and purpose and be present in the body.
  On another day, participants completed 30 min of Quiet Rest
Arm/Group | YogaFit | Quiet Rest
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No